CLINICAL TRIAL: NCT06995963
Title: Impact of TURP on Quality of Life in Patients With Benign Prostatic Hyperplasia: A Retrospective Study
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Gonesse (Other)
Responsible Party: Sponsor
Other Study IDs: 0099_UROLOGIE
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Prostatic Hyperplasia; Prostatectomy; Transurethral Resection of Prostate; Quality of Life; Urinary Tract Symptoms; Treatment Outcome
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study looks at how a common surgery called TURP (Transurethral Resection of the Prostate) affects the quality of life in men with benign prostatic hyperplasia (BPH), a non-cancerous enlargement of the prostate. By reviewing past medical records of patients who had this surgery, researchers will evaluate how urinary symptoms and overall well-being changed after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Male patients with urinary symptoms related to prostatic obstruction
* Patients who underwent transurethral resection of the prostate (TURP)
* Availability of pre- and post-operative data (including IPSS)

Exclusion Criteria:

* Patients with urinary symptoms not related to prostatic obstruction
* Patients who did not undergo TURP
* Incomplete or missing clinical data required for analysis

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of adult male patients diagnosed with benign prostatic hyperplasia (BPH) who underwent transurethral resection of the prostate (TURP) at a single medical center. Participants will be selected retrospectively from medical records of patients treated between February and April. All included patients must have urinary symptoms related to prostatic obstruction and complete pre- and post-operative data available, including IPSS scores.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Change in urinary symptoms after TURP, measured by the IPSS | From baseline (pre-surgery) to 1-3 months post-surgery

CONTACTS AND LOCATIONS:
Locations (1):
- France, Gonesse, France, France